CLINICAL TRIAL: NCT01474733
Title: Effects of a Longitudinal Health Literacy Training Program on Family Medicine Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Cliff Coleman, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: OHSU IRB#00008039
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Health Literacy
Keywords: resident education; health literacy; curriculum
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- educational intervention (Experimental): participants undergo a series of educational interventions over 3 years
  Interventions: Other: educational intervention

INTERVENTIONS:
Other: educational intervention — series of lectures and workshops on health literacy

SUMMARY:
1. Briefly describe the purpose of this protocol: This study is designed to evaluate the effectiveness of an educational training program on the topic of health literacy for Family Medicine residents. The hypothesis being tested is that training residents about health literacy will result in improvements in residents' knowledge, skills, and attitudes with respect to health literacy.
2. Briefly summarize how participants are recruited: OHSU Family Medicine Interns attending mandatory trainings on the topic of health literacy throughout the three years of the residency program will be invited to participate in the study.
3. Briefly describe the procedures subjects will undergo: Completion of a short self-administered anonymous survey before and after a variety of learning sessions on the topic of health literacy.
4. If applicable, briefly describe survey/interview instruments used: A 12-item pre-test questionnaire and 13-item post-test questionnaire designed to assess individuals' knowledge about health literacy, and intended clinical practices with respect to health literacy.
5. If this is a clinical trial using an experimental drug and/or device, or an approved drug and/or device used for an unapproved purpose, briefly describe the drug and/or device: n/a
6. Briefly describe how the data will be analyzed to address the purpose of the protocol: Demographics and responses to individual items will be reported as frequencies and percentages within the sample. We will use a chi-square analysis to stratify responses by demographic groups and t-tests to measure possible changes over time

ELIGIBILITY:
Inclusion Criteria:

-Family medicine resident entering in summer 2011 at OHSU Department of Family Medicine

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
knowledge about health literacy | 3 years
  as measured by a standardized questionnaire

SECONDARY OUTCOMES:
clear communication skills | 3 years
  As measured by performance on an OSCE

CONTACTS AND LOCATIONS:
Overall Officials: Clifford A Coleman, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU Richmond Clinic, Portland, Oregon, United States